CLINICAL TRIAL: NCT01979536
Title: A Randomized Phase 2 Trial of Brentuximab Vedotin (SGN35, NSC# 749710), or Crizotinib (NSC#749005, Commercially Labeled) in Combination With Chemotherapy for Newly Diagnosed Patients With Anaplastic Large Cell Lymphoma (ALCL)
Brief Title: Brentuximab Vedotin or Crizotinib and Combination Chemotherapy in Treating Patients With Newly Diagnosed Stage II-IV Anaplastic Large Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02167; NCI-2013-02167 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s14-01970; COG-ANHL12P1; ANHL12P1 (Other: Children's Oncology Group); ANHL12P1 (Other: CTEP); U10CA098543 (NIH); U10CA180886 (NIH)
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Results first posted 2022-07-06 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Positive; Ann Arbor Stage II Noncutaneous Childhood Anaplastic Large Cell Lymphoma; Ann Arbor Stage III Noncutaneous Childhood Anaplastic Large Cell Lymphoma; Ann Arbor Stage IV Noncutaneous Childhood Anaplastic Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic | interventions — Brentuximab Vedotin; Crizotinib; Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Etoposide; Ifosfamide; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm BV (brentuximab vedotin, combination chemotherapy) (Experimental): COURSE A (CYCLES 1, 3, AND 5): Patients receive brentuximab vedotin IV over 30 minutes on day 1, dexamethasone PO BID or IV on days 1-5, ifosfamide IV over 60 minutes on days 1-5, methotrexate IV over 3 hours on day 1, cytarabine IV over 1-30 minutes every 12 hours for 4 doses on days 4 and 5, and etoposide IV over 2 hours on days 4 and 5.
  COURSE B (CYCLES 2, 4, AND 6): Patients receive brentuximab vedotin, dexamethasone, and methotrexate as in Arm BV, Course A. Patients also receive cyclophosphamide IV over 15-30 minutes on days 1-5 and doxorubicin hydrochloride IV over 1-15 minutes on days 4 and 5.
  Interventions: Drug: Brentuximab Vedotin; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate
- Arm CZ (crizotinib, combination chemotherapy) (Experimental): COURSE A (CYCLES 1, 3, AND 5): Patients receive crizotinib PO BID on days 1-21 and dexamethasone, ifosfamide, methotrexate, cytarabine, and etoposide as in Arm BV, Course A.
  COURSE B (CYCLES 2, 4, AND 6): Patients receive crizotinib PO BID as in Arm CZ, Course A and dexamethasone, cyclophosphamide, methotrexate, and doxorubicin hydrochloride as in Arm BV, Course B.
  Interventions: Drug: Crizotinib; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
  Arms: Arm BV (brentuximab vedotin, combination chemotherapy)
Drug: Crizotinib — Given PO
  Other Names: MET Tyrosine Kinase Inhibitor PF-02341066; PF-02341066; PF-2341066; PF02341066; Xalkori
  Arms: Arm CZ (crizotinib, combination chemotherapy)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B-518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719; WR-138719
Drug: Cytarabine — Given IT and IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP16
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Drug: Methotrexate — Given IT and IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039

SUMMARY:
This partially randomized phase II trial studies how well brentuximab vedotin or crizotinib and combination chemotherapy works in treating patients with newly diagnosed stage II-IV anaplastic large cell lymphoma. Brentuximab vedotin is a monoclonal antibody, called brentuximab, linked to a toxic agent called vedotin. Brentuximab attaches to CD30 positive cancer cells in targeted way and delivers vedotin to kill them. Crizotinib and methotrexate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether brentuximab vedotin and combination chemotherapy is more effective than crizotinib and combination chemotherapy in treating anaplastic large cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the tolerability of brentuximab vedotin given in combination with standard chemotherapy (anaplastic large cell lymphoma [ALCL]99) and to determine the tolerability of crizotinib given in combination with chemotherapy (ALCL99).

II. To estimate the event free survival (EFS) of Arm brentuximab vedotin (BV) and Arm crizotinib (CZ) and contrast these to historical control data.

SECONDARY OBJECTIVES:

I. To determine the prognostic significance of minimal disseminated disease (MDD) at diagnosis and minimal residual disease (MRD) as measured by real-time (RT)-polymerase chain reaction (PCR) in peripheral blood.

OUTLINE: Patients with body surface area (BSA) < 0.9 m^2 were non-randomly assigned to Arm BV while it was open and were not eligible for the trial while Arm BV was closed. Patients with BSA >= 0.9 m^2 were randomly assigned 1:1 to Arm BV or Arm CZ while both were open and were non-randomly assigned to the open arm while only one of the two arms was open.

ARM BV:

COURSE A (CYCLES 1, 3, AND 5): Patients receive brentuximab vedotin (1.8 mg/dg/dose - Max dose 180 mg) intravenously (IV) over 30 minutes on day 1, dexamethasone orally (PO) twice daily (BID) or IV on days 1-5, ifosfamide IV over 60 minutes on days 1-5, methotrexate IV over 3 hours on day 1, cytarabine IV over 1-30 minutes every 12 hours for 4 doses on days 4 and 5, and etoposide IV over 2 hours on days 4 and 5.

COURSE B (CYCLES 2, 4, AND 6): Patients receive brentuximab vedotin (1.8 mg/dg/dose - Max dose 180 mg), dexamethasone, and methotrexate as in Arm BV, Course A. Patients also receive cyclophosphamide IV over 15-30 minutes on days 1-5 and doxorubicin hydrochloride IV over 1-15 minutes on days 4 and 5.

ARM CZ:

COURSE A (CYCLES 1, 3, AND 5): Patients receive crizotinib (165 mg/m^2) PO BID on days 1-21 and dexamethasone, ifosfamide, methotrexate, cytarabine, and etoposide as in Arm BV, Course A.

COURSE B (CYCLES 2, 4, AND 6): Patients receive crizotinib (165 mg/m^2) PO BID as in Arm CZ, Course A and dexamethasone, cyclophosphamide, methotrexate, and doxorubicin hydrochloride as in Arm BV, Course B.

In all arms, treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, 9, 12, 18, 24, 36, 48, and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with histologically proven ALCL (International Classification of Diseases for Oncology [ICD-0] code: 9714/3)
* Disease must be cluster of differentiation (CD)30 positive
* Disease must be anaplastic lymphoma kinase (ALK) positive (defined by local institutional standards)
* Patients must have stage II, III, or IV disease
* Patients must have a life expectancy of >= 8 weeks
* Adequate Liver Function Defined As:
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x upper limit of normal (ULN) for age; for the purpose of this study, the ULN for ALT is 45 U/L (within 7 days prior to enrollment)
* If the lab abnormality is thought to be due to the lymphoma the patient is eligible and dose adjustments should be made
* Adequate Cardiac Function Defined As:
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by radionuclide angiogram
* Adequate Pulmonary Function Defined As:
* Patients with a history of pulmonary dysfunction must have no evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and a pulse oximetry > 92% while breathing room air unless current dysfunction is due to the lymphoma in which case the patient is eligible

Exclusion Criteria:

* Patients with central nervous system (CNS) disease are not eligible
* Patients with disease limited to the skin are not eligible, regardless of how wide-spread
* Patients with stage I disease are not eligible
* Patients who have received any prior cytotoxic chemotherapy for the current diagnosis of ALCL or any cancer diagnosed previously are not eligible
* Previous steroid treatment and/or radiation treatment is not allowed unless it is for the emergent management of a mediastinal mass; emergent steroid treatment and/or radiation treatment should stop once protocol therapy is initiated
* Intrathecal chemotherapy prior to enrollment is allowed for the current diagnosis of ALCL as long as adequate cerebrospinal fluid (CSF) is obtained prior to administration of the intrathecal chemotherapy and subsequently demonstrated to be negative for ALCL
* Female patients who are pregnant are not eligible; pregnancy tests must be obtained in girls who are post menarchal
* Lactating females are not eligible unless they have agreed not to breastfeed their infants
* Sexually active patients of reproductive potential are not eligible unless they agree to use an effective contraceptive method for the duration of treatment and for 3 months after stopping treatment
* Patients with Down syndrome are not eligible due to the amount of methotrexate and potential for side effects
* Patients with an immunodeficiency that existed prior to diagnosis such as primary immunodeficiency syndromes or organ transplant recipients are not eligible
* Cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) substrates with narrow therapeutic indices: Patients chronically receiving medications known to be metabolized by CYP3A4 and with narrow therapeutic indices including pimozide, aripiprazole, triazolam, ergotamine and halofantrine are not eligible; the topical use of these medications (if applicable) is allowed
* CYP3A4 inhibitors: patients chronically receiving drugs that are known potent CYP3A4 inhibitors within 7 days prior to study enrollment, including but not limited to ketoconazole, itraconazole, clarithromycin, erythromycin, ritonavir, indinavir, nelfinavir, saquinavir, delavirdine, nefazodone, diltiazem, verapamil, and grapefruit juice are not eligible; the topical use of these medications (if applicable), e.g. 2% ketoconazole cream, is allowed
* CYP3A4 inducers: patients chronically receiving drugs that are known potent CYP3A4 inducers within 12 days prior to study enrollment, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, ritonavir, and St. John's wort are not eligible; the topical use of these medications (if applicable) is allowed
* Patients that are known to be positive for human immunodeficiency virus (HIV) are not eligible; note: inclusion of HIV positive patients will be considered at a later date
* Patients who weigh < 10 kg are not eligible

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2013-11-13 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Lowe, Principal Investigator — Children's Oncology Group
Locations (154):
- United States (154):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Beaumont Children's Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Lowe EJ, Reilly AF, Lim MS, Gross TG, Saguilig L, Barkauskas DA, Wu R, Alexander S, Bollard CM. Crizotinib in Combination With Chemotherapy for Pediatric Patients With ALK+ Anaplastic Large-Cell Lymphoma: The Results of Children's Oncology Group Trial ANHL12P1. J Clin Oncol. 2023 Apr 10;41(11):2043-2053. doi: 10.1200/JCO.22.00272. Epub 2022 Dec 19. PMID 36534942
- [Derived] Lowe EJ, Reilly AF, Lim MS, Gross TG, Saguilig L, Barkauskas DA, Wu R, Alexander S, Bollard CM. Brentuximab vedotin in combination with chemotherapy for pediatric patients with ALK+ ALCL: results of COG trial ANHL12P1. Blood. 2021 Jul 1;137(26):3595-3603. doi: 10.1182/blood.2020009806. PMID 33684925

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm BV (Brentuximab Vedotin, Combination Chemotherapy): COURSE A (CYCLES 1, 3, AND 5): Patients receive brentuximab vedotin IV over 30 minutes on day 1, dexamethasone PO BID or IV on days 1-5, ifosfamide IV over 60 minutes on days 1-5, methotrexate IV over 3 hours on day 1, cytarabine IV over 1-30 minutes every 12 hours for 4 doses on days 4 and 5, and etoposide IV over 2 hours on days 4 and 5.
  COURSE B (CYCLES 2, 4, AND 6): Patients receive brentuximab vedotin, dexamethasone, and methotrexate as in Arm BV, Course A. Patients also receive cyclophosphamide IV over 15-30 minutes on days 1-5 and doxorubicin hydrochloride IV over 1-15 minutes on days 4 and 5.
  Brentuximab Vedotin: Given IV
  Cyclophosphamide: Given IV
  Cytarabine: Given IT and IV
  Dexamethasone: Given PO or IV
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Methotrexate: Given IT and IV
- Arm CZ (Crizotinib, Combination Chemotherapy): COURSE A (CYCLES 1, 3, AND 5): Patients receive crizotinib PO BID on days 1-21 and dexamethasone, ifosfamide, methotrexate, cytarabine, and etoposide as in Arm BV, Course A.
  COURSE B (CYCLES 2, 4, AND 6): Patients receive crizotinib as in Arm CZ, Course A and dexamethasone, cyclophosphamide, methotrexate, and doxorubicin hydrochloride as in Arm BV, Course B.
  Crizotinib: Given PO
  Cyclophosphamide: Given IV
  Cytarabine: Given IT and IV
  Dexamethasone: Given PO or IV
  Doxorubicin Hydrochloride: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Methotrexate: Given IT and IV
Period: Overall Study
Arm/Group | Arm BV (Brentuximab Vedotin, Combination Chemotherapy) | Arm CZ (Crizotinib, Combination Chemotherapy)
Started | 68 | 69
Completed | 66 | 61
Not Completed | 2 | 8
Not completed — Physician Decision | 2 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Refusal | 0 | 1
Not completed — Relapse | 0 | 1
Not completed — Study terminated by Sponsor | 0 | 1
Not completed — Did not start treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm BV (Brentuximab Vedotin, Combination Chemotherapy) | Arm CZ (Crizotinib, Combination Chemotherapy) | Total
Number analyzed (Participants) | 68 | 69 | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64 | 65 | 129
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (4.9) | 13.6 (3.3) | 12.2 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 43 | 47 | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 10 | 15
  Not Hispanic or Latino | 60 | 56 | 116
  Unknown or Not Reported | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 14 | 22
  White | 48 | 46 | 94
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 68 | 69 | 137

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Grade 3+ Non-hematologic Adverse Events
Description: Will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Toxicities will be summarized by individual toxicity counts separated by arm.
Time Frame: Up to 60 months
Population: 1 Arm BV patient who did not receive at least one dose of brentuximab vedotin and 3 Arm CZ patients who did not receive at least one dose of crizotinib are excluded from these analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm BV (Brentuximab Vedotin, Combination Chemotherapy) | Arm CZ (Crizotinib, Combination Chemotherapy)
Number analyzed (Participants) | 67 | 66
Percentage of patients | 80.6 [69.1 to 89.2] | 87.9 [77.5 to 94.6]

2. Primary Outcome: Event Free Survival (EFS)
Description: The Kaplan-Meier method will be used to estimate the 2-year EFS for each of the treatment regimens.
Time Frame: Time from study entry until progressive disease, relapse, or death, assessed up to 2 years
Population: 1 Arm CZ patient who did not start treatment is excluded from analyses of EFS.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm BV (Brentuximab Vedotin, Combination Chemotherapy) | Arm CZ (Crizotinib, Combination Chemotherapy)
Number analyzed (Participants) | 68 | 68
Percentage of patients | 78.8 [67.2 to 87.1] | 76.8 [68.5 to 88.1]

3. Secondary Outcome: Prognostic Significance of Minimal Residual Disease
Description: Analyzed by estimating the 2-year EFS of negative MRD and positive MRD by arm. Minimal disease was performed using serial assessments of the t(2;5)(p23;q35) NPM-ALK fusion transcript using quantitative RT-PCR. Quantitative RT-PCR was performed by extracting total RNA from peripheral blood specimens. Peripheral blood samples were obtained at baseline, on day 1 of cycle 1, and on day 1 of cycle 2. The normalized copy numbers (NCN) were expressed as copy numbers of NPM-ALK per 104 copies of ABL. Minimal disease (MDD) was defined as >10 NCN at baseline.
Time Frame: Baseline up to progressive disease, relapse, or death, assessed up to 2 years
Population: 11 Arm BV patients without adequate MDD baseline data, 1 Arm CZ patient who did not start treatment, and 11 Arm CZ patients without adequate MDD baseline data are excluded from these analyses.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- MRD Negative Arm BV (Brentuximab Vedotin, Combination Chemotherapy); MRD Positive Arm BV (Brentuximab Vedotin, Combination Chemotherapy): COURSE A (CYCLES 1, 3, AND 5): Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1, dexamethasone orally (PO) twice daily (BID) or IV on days 1-5, ifosfamide IV over 60 minutes on days 1-5, methotrexate IV over 3 hours on day 1, cytarabine IV over 1-30 minutes every 12 hours for 4 doses on days 4 and 5, and etoposide IV over 2 hours on days 4 and 5.
  COURSE B (CYCLES 2, 4, AND 6): Patients receive brentuximab vedotin, dexamethasone, and methotrexate as in Arm BV, Course A. Patients also receive cyclophosphamide IV over 15-30 minutes on days 1-5 and doxorubicin hydrochloride IV over 1-15 minutes on days 4 and 5.
- MRD Negative Arm CZ (Crizotinib, Combination Chemotherapy); MRD Positive Arm CZ (Crizotinib, Combination Chemotherapy): COURSE A (CYCLES 1, 3, AND 5): Patients receive crizotinib PO BID on days 1-21 and dexamethasone, ifosfamide, methotrexate, cytarabine, and etoposide as in Arm BV, Course A.
  COURSE B (CYCLES 2, 4, AND 6): Patients receive crizotinib as in Arm CZ, Course A and dexamethasone, cyclophosphamide, methotrexate, and doxorubicin hydrochloride as in Arm BV, Course B.
Arm/Group | MRD Negative Arm BV (Brentuximab Vedotin, Combination Chemotherapy) | MRD Positive Arm BV (Brentuximab Vedotin, Combination Chemotherapy) | MRD Negative Arm CZ (Crizotinib, Combination Chemotherapy) | MRD Positive Arm CZ (Crizotinib, Combination Chemotherapy)
Number analyzed (Participants) | 38 | 19 | 37 | 20
Percentage of patients | 89 [73.1 to 95.7] | 52.6 [28.7 to 71.9] | 85.6 [68.6 to 93.8] | 58.1 [33.4 to 76.4]

ADVERSE EVENTS:
Time Frame: Enrollment up to 5 years after enrollment
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Patients who did not start treatment are excluded from reporting of AEs. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Arm BV (Brentuximab Vedotin, Combination Chemotherapy) | Arm CZ (Crizotinib, Combination Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 3/68 | 3/68
Serious Adverse Events (participants affected / at risk) | 24/68 | 41/68
Other Adverse Events (participants affected / at risk) | 57/68 | 55/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm BV (Brentuximab Vedotin, Combination Chemotherapy) (N=68) | Arm CZ (Crizotinib, Combination Chemotherapy) (N=68)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 7
Sinus tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 12 | 16
Nausea (Gastrointestinal disorders) | 0 | 2
Oral pain (Gastrointestinal disorders) | 3 | 1
Typhlitis (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3
Death NOS (General disorders) | 1 | 3
Fever (General disorders) | 2 | 2
Anaphylaxis (Immune system disorders) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 1 | 3
Skin infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 5 | 3
Blood bilirubin increased (Investigations) | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 2 | 0
White blood cell decreased (Investigations) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 5
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Tracheal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 3
Thromboembolic event (Vascular disorders) | 4 | 13 — Only Arm CZ was stopped due to toxicity (thromboembolic events). The high rate of thromboembolic events could be secondary to chance or a result of crizotinib in combination with this specific chemotherapy.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm BV (Brentuximab Vedotin, Combination Chemotherapy) (N=68) | Arm CZ (Crizotinib, Combination Chemotherapy) (N=68)
Anemia (Blood and lymphatic system disorders) | 22 | 27
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 30 | 30
Periorbital edema (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 6 | 11
Nausea (Gastrointestinal disorders) | 1 | 2
Oral pain (Gastrointestinal disorders) | 1 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 1
Endocarditis infective (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 8 | 5
Kidney infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 3 | 1
Otitis media (Infections and infestations) | 0 | 1
Scrotal infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 9 | 9
Alkaline phosphatase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 3
Creatinine increased (Investigations) | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1
Fibrinogen decreased (Investigations) | 0 | 1
GGT increased (Investigations) | 0 | 3
Lymphocyte count decreased (Investigations) | 17 | 18
Lymphocyte count increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 26 | 32
Platelet count decreased (Investigations) | 21 | 26
Weight gain (Investigations) | 0 | 1
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 17 | 25
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalemia (Metabolism and nutrition disorders) | 9 | 10
Hyponatremia (Metabolism and nutrition disorders) | 5 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/36/NCT01979536/Prot_SAP_000.pdf